CLINICAL TRIAL: NCT01554839
Title: The Family of Heroes Program for Veterans and Their Families: An Evaluation of an Online Educational Tool for Helping Veterans.
Brief Title: The Family of Heroes: an Evaluation of an Online Educational Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Veterans Affairs, New Jersey (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alejandro Interian, PhD, Clinical Psychologist, Department of Veterans Affairs, New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIRB#01165
Record Dates: First submitted 2012-03-05; First posted 2012-03-15 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2013-06

CONDITIONS: Post Traumatic Stress Disorder; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — BaseLine dental cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): Treatment group participates in 1 hour online educational tool in addition to baseline and follow up surveys
  Interventions: Behavioral: "Family of Heroes"; Behavioral: Baseline and Follow up Surveys
- Non Treatment Group (Placebo Comparator): Non Treatment group participates in baseline and follow up surveys
  Interventions: Behavioral: Baseline and Follow up Surveys

INTERVENTIONS:
Behavioral: "Family of Heroes" — One hour online educational tool
  Arms: Treatment Group
Behavioral: Baseline and Follow up Surveys — Baseline and follow up questionaires completed online

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a unique web based educational tool called "Family of Heroes," which is designed to educate families about Post Traumatic Stress Disorder (PTSD) and provide them with practical tools for interacting with affected veteran family members. The study includes veterans and a family member of their choosing. Participants are randomly assigned to a group which takes the online training or a group that does not take the training. Both groups complete a baseline questionnaire and a follow up questionaire 60 days later. The study will examine the number of Veteran Affairs (VA) mental health visits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Operation Iraqi Freedom/ Operation Enduring Freedom (OIF/OEF) veteran
* Positive for PTSD, based on PTSD Checklist (PCL) score greater than or equal to 50
* Availability of a family member who is both willing to participate in the study AND has contact with the veteran 3 or more times per week
* Ability to access a computer with internet access to take educational training and surveys

Exclusion Criteria:

* Not and OIF/OEF veteran
* Negative for PTSD, based on PCL score less than 50
* Unavailability of a family member who is both willing to participate in the study or has contact with the veteran 3 or more times per week
* Inability to access a computer with internet access to take the educational training and surveys

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Mental Health Treatment Engagement | 6 months post enrollment
  Number of mental health visits attended. Obtained from chart review.

SECONDARY OUTCOMES:
Change in Perceived Criticism Score | Baseline and 2 months
  4 questions answered on a scale of 1 to 10; 1 being not at all critical and 10 being very critical.
Change in Family Empowerment Scale Score | Baseline and 2 months
  12 questions answered on a scale of 1 through 5. 1 = not true at all, 2 = mostly not true, 3 = somewhat true, 4 = mostly true, and 5 = very true.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Interian, PhD, Principal Investigator — Department of Veteran Affairs, New Jersey
Locations (1):
- VANJHCS (Veterans Administration New Jersey Health Care Services), Lyons, New Jersey, United States

REFERENCES:
- [Derived] Interian A, Kline A, Perlick D, Dixon L, Feder A, Weiner MD, Goldstein MF, Hennessy K, St Hill L, Losonczy M. Randomized controlled trial of a brief Internet-based intervention for families of Veterans with posttraumatic stress disorder. J Rehabil Res Dev. 2016;53(5):629-640. doi: 10.1682/JRRD.2014.10.0257. PMID 27898154